CLINICAL TRIAL: NCT02272465
Title: Prehospital Resuscitation On Helicopter Study
Acronym: PROHS
Status: Completed | Type: Observational
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: University of Cincinnati (Other); Mayo Clinic (Other); Oregon Health and Science University (Other); University of Washington (Other); University of Maryland (Other); University of Alabama at Birmingham (Other); University of Arizona (Other); University of Southern California (Other); National Heart, Lung, and Blood Institute (NHLBI) (NIH); Resuscitation Outcomes Consortium (Network)
Responsible Party: Principal Investigator, John Holcomb, M.D., Chief Division of Acute Care Surgery, Director Center for Translational Injury Research, The University of Texas Health Science Center, Houston
Other Study IDs: HSC-GEN-14-0735; U01HL077863 (NIH)
Record Dates: First submitted 2014-10-09; First posted 2014-10-23 (Estimated); Last update posted 2015-12-08 (Estimated); Status verified 2015-12

CONDITIONS: Traumatic Injuries
Keywords: pre-hospital resuscitation, helicopter, trauma
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Received blood products during transport: There is no intervention as this is an observational study. The first group will be the patients that received blood products during the helicopter transport from the scene of the injury per standard of care guidelines at the participating institutions.
  Interventions: Other: No intervention
- Received crystalloid during transport: There is no study intervention. The second group will be the patients that did not receive blood products during the helicopter transport because blood products are not available or part of the standard of care during flight.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Observational study

SUMMARY:
The Prehospital Resuscitation On Helicopter Study (PROHS) is a pragmatic, multicenter, prospective observational study of air ambulance-based prehospital resuscitation regimens currently utilized at the participating sites. Patients will be enrolled at participating sites that currently have blood products available on air ambulances and other sites that do not. This study will not change the current prehospital standard of care for resuscitation. The primary outcome will be in-hospital mortality and the primary unit of analysis will be the patient. Other outcomes of interest will include time to hemostasis, hospital length-of-stay, number of ventilator-free and ICU-free days, incidence of major surgical procedures, complications (transfusion-related acute lung injury [TRALI], acute kidney injury [AKI], multiple organ failure [MOF], acute respiratory distress syndrome [ARDS], sepsis, intra-abdominal complications, thromboembolic complications, compartment syndromes), lifesaving interventions, the amount and type of blood products and concentrates transfused (including prehospital), wastage of prehospital blood products and concentrates, use of external and internal hemostatic devices, and functional status at discharge/discharge destination.

DETAILED DESCRIPTION:
All patients arriving to the participating center's trauma emergency department via helicopter directly from the scene will be screened and initial data collected. Of that group, all patients who meet the "highest risk" category (based on vital signs, type of injury, use of tourniquet, and/or intubation) or received blood during transport will be followed through "direct observation" through the initial resuscitation period and then indirectly through medical chart review until hospital discharge or 30 days after admission (whichever occurs first).

ELIGIBILITY:
Inclusion Criteria:

Criteria for "at risk" population

* Patients with traumatic injuries received directly from the scene via air ambulance service (did not receive a lifesaving intervention at an outside hospital or healthcare facility)
* Estimated age of 15 or older or greater than/equal to a weight of 50 kg, if age unknown Criteria for "highest risk" population
* Meet at least one of the following during prehospital care: HR >120 bpm, SBP ≤90 mmHg, penetrating truncal injury, tourniquet application, pelvic binder application or intubation.
* Received blood products during transport (for those facilities with blood product availability)

Exclusion Criteria:

* Prisoners (defined as those received directly from a correctional facility.

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target population for this study is trauma patients who are transported to one of the participating Level I trauma centers via air ambulance, directly from the scene, and meet the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 1049 (Actual)
Dates: Start 2015-01; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
In-patient mortality. | Up to 30 days

OTHER OUTCOMES:
Length of hospital stay | Up to 30 days
  The total # of hospital days
Number of ICU days | Up to 30 days
Number of Ventilator days | Up to 30 days
Blood product usage | Up to 30 days
  Number of RBCs, plasma and platelets used during resuscitation.
GOSE score | Up to 30 days
  GOSE score to measure functional status at time of discharge
Number of patients with complications | Up to 30 days
  Will evaluate the number of patients who experienced common complication following traumatic injury.
Number of patients who required hemostatic devices | up to 30 days
  The use of external and internal hemostatic devices.

CONTACTS AND LOCATIONS:
Overall Officials: John Holcomb, M.D., Principal Investigator — The University of Texas Health Science Center, Houston
Locations (9):
- United States (9):
  - University of Alabama, Birmingham, Alabama
  - University of Arizona, Tucson, Arizona
  - University of Southern California, Los Angeles, Los Angeles, California
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Mayo Medical Center, Rochester, Minnesota
  - University of Cincinnati, Cincinnati, Ohio
  - Oregon Health and Science University, Portland, Oregon
  - Memorial Hermann Hospital - Texas Medical Center, Houston, Texas
  - University of Washington- Harborview Medical Center, Seattle, Washington